CLINICAL TRIAL: NCT00295867
Title: Pilot Study to Evaluate the Effect of Zoledronic Acid (Zometa) on Occult Malignant Bone Marrow Cells in Patients With High Risk Early Stage Breast Cancer
Brief Title: Zoledronate in Treating Bone Marrow Micrometastases in Women With Stage I, Stage II, or Stage III Breast Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of California, San Francisco (Other)
Collaborators: Novartis (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 037519; UCSF-H6961-24352-02 (Other: University of California, San Francisco); 10-01674 (Other: University of California, San Francisco)
Record Dates: First submitted 2006-02-23; First posted 2006-02-24 (Estimated); Results first posted 2020-05-12 (Actual); Last update posted 2020-05-12 (Actual); Status verified 2020-05

CONDITIONS: Breast Cancer
Keywords: stage I breast cancer; stage II breast cancer; stage IIIA breast cancer; stage IIIB breast cancer; stage IIIC breast cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — Zoledronic Acid

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Zoledronic Acid (Experimental): Patients women with early stage breast cancer and evidence of occult malignant cells in bone marrow aspirates following adjuvant chemotherapy will receive zoledronic acid (Zometa) 4mg, given intravenously over 15 minutes, once a month for two years.
  Interventions: Drug: Zoledronic Acid

INTERVENTIONS:
Drug: Zoledronic Acid — Zoledronic acid is a new, highly potent, heterocyclic nitrogen-containing third generation bisphosphonate that has demonstrated 40- to 850- fold greater potency than pamidronate in preclinical models of bone resorption. The mechanism of action of nitrogen-containing bisphosphonates such as pamidronate and zoledronic acid appears to involve inhibition of the mevalonate pathway
  Other Names: Zometa; Zoledronate

SUMMARY:
RATIONALE: Zoledronate may delay or prevent bone marrow metastases in patients with breast cancer.

PURPOSE: This phase II trial is studying how well zoledronate works in treating bone marrow micrometastases in women with stage I, stage II, or stage III breast cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* Determine the response of bone marrow micrometastases, as measured by immunocytochemistry/flow cytometry (IC/FC), during and after 2 years of treatment with zoledronate in women with stage I-III breast cancer.

Secondary

* Evaluate the effects of zoledronate on the bone osteoclast activation marker, n-telopeptide, in these patients.
* Evaluate the incidence of distant recurrences in high-risk women with early-stage breast cancer and bone marrow micrometastases who receive adjuvant zoledronate.

OUTLINE: This is a pilot study.

Patients receive zoledronate IV over 15 minutes once a month for 2 years in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed every 6 months.

PROJECTED ACCRUAL: A total of 35 patients will be accrued for this study.

ELIGIBILITY:
Inclusion Criteria

1. Women > 18 years of age with histologically or cytologically confirmed stage I, II or III breast cancer.
2. If adjuvant chemotherapy is recommended, it must be completed before study start.
3. Bone marrow aspirate positive by IC/FC assay

   a. Definition of positive: > 4 MM/ml b. Timing of bone marrow aspiration to determine study eligibility: i. If patient is to receive either no adjuvant therapy or hormonal therapy alone, the aspiration may be performed at diagnosis as part of the large MM study at University of California, San Francisco, or following diagnosis if the patient received initial surgery elsewhere. This is also true for patients who have surgery following neoadjuvant therapy for breast cancer.

   ii. If the patient is to receive adjuvant chemotherapy, the aspiration will be performed at least three weeks after chemotherapy has been completed.
4. Adequate renal function as defined by:

   a. Creatinine must be < upper limit of normal
5. Normal liver function tests including total bilirubin, alkaline phosphatase, and aspartate aminotransferase (AST) / serum glutamic-oxaloacetic transaminase (SGOT)
6. Ability to understand and sign informed consent.
7. Concomitant hormonal therapy is allowed
8. Concomitant radiation therapy is allowed
9. Patients who have had surgery following neoadjuvant chemotherapy or hormonal therapy are eligible to participate in this trial

Exclusion Criteria

1. History of allergy to bisphosphonates. Acute phase reactions occur in up to 24% of patients and disappear with subsequent dosing. An acute phase reaction does not qualify as an allergic reaction.
2. History of renal insufficiency. Renal insufficiency is defined by a serum creatinine greater than the upper limit of normal or a creatinine clearance < 50 mL/min due to any underlying cause.
3. Karnofsky Performance status < 90%.
4. Any significant medical condition that might interfere with treatment.
5. Women participating in this study are not allowed to receive other bisphosphonate therapy during the study period, either oral or intravenous.
6. Patients who are pregnant

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 45 (Actual)
Dates: Start 2004-11-03 (Actual); Primary Completion 2011-06 (Actual); Study Completion 2013-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Hope S. Rugo, MD, Principal Investigator — University of California, San Francisco
Locations (1):
- University of California, San Francisco, San Francisco, California, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Adams A, Jakob T, Huth A, Monsef I, Ernst M, Kopp M, Caro-Valenzuela J, Wockel A, Skoetz N. Bone-modifying agents for reducing bone loss in women with early and locally advanced breast cancer: a network meta-analysis. Cochrane Database Syst Rev. 2024 Jul 9;7(7):CD013451. doi: 10.1002/14651858.CD013451.pub2. PMID 38979716

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Patients were enrolled between October 2004 and October 2007. Patients were recruited in a medical clinic at the University of California, San Francisco Helen Diller Family Comprehensive Cancer Center.
Groups:
- Zoledronic Acid: Patients who had greater than 4 disseminated tumor cells (DTCs)/mL present following neoadjuvant or adjuvant chemotherapy for early stage breast cancer were treated with 4mg zoledronic acid each month for 24 months.
Period: Overall Study
Arm/Group | Zoledronic Acid
Started | 45
Completed | 34
Not Completed | 11

BASELINE CHARACTERISTICS:
Arm/Group | Zoledronic Acid
Number analyzed (Participants) | 45
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 45
  >=65 years | 0
Age, Continuous [Mean (Full Range); unit: years] | 46 [29 to 64]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 45
  Male | 0
Region of Enrollment [Number; unit: participants]
  United States | 45

OUTCOME MEASURES:

1. Primary Outcome: Response of Bone Marrow Micrometastases
Description: Median change in disseminated tumor cells (DTCs)/mL from baseline after 24 months
Time Frame: up to 2 years
Population: Only 34 patients had bone marrow aspiration (BMA) at 24 mos required for this analysis
Measure: Median (Full Range); unit: DTCs/mL
Arm/Group | Zoledronic Acid
Number analyzed (Participants) | 34
DTCs/mL | -4.5 [-5.9 to 43.1]

2. Secondary Outcome: Change in N-telopeptide Level
Description: N-telopeptide levels in urine will be recorded to evaluate the effect of zoledronic acid on bone mineralization (nmol bone collagen equivalents/mmol creatinine) at baseline and after 24 months on study treatment
Time Frame: up to 2 years
Population: N-telopeptide levels in urine data not collected
Arm/Group | Zoledronic Acid
Number analyzed (Participants) | 0

3. Secondary Outcome: Number of Patients With Incidences of Distant Recurrence
Description: Distant breast cancer recurrence is when the cancer has spread to another organ within the body.
Time Frame: up to 5 years post initiation of treatment
Measure: Number; unit: participants
Arm/Group | Zoledronic Acid
Number analyzed (Participants) | 34
participants | 6

ADVERSE EVENTS:
Time Frame: Two years
Arm/Group | Zoledronic Acid
All-Cause Mortality (participants affected / at risk) | 2/45
Serious Adverse Events (participants affected / at risk) | 1/45
Other Adverse Events (participants affected / at risk) | 33/45
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Zoledronic Acid (N=45)
appendicitis (Gastrointestinal disorders) | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Zoledronic Acid (N=45)
Myalgia (Musculoskeletal and connective tissue disorders) | 18
Back pain (Musculoskeletal and connective tissue disorders) | 2
Bone pain (Musculoskeletal and connective tissue disorders) | 4
Cough (Respiratory, thoracic and mediastinal disorders) | 1
Fatigue (General disorders) | 14
Fever (General disorders) | 5
Flu like symptoms (General disorders) | 10
grinding teeth (Gastrointestinal disorders) | 1
Headache (Nervous system disorders) | 1
Hip pain (Musculoskeletal and connective tissue disorders) | 1
Creatinine increased (Investigations) | 1
Jaw pain (Musculoskeletal and connective tissue disorders) | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 2
Lightheadedness (Nervous system disorders) | 2
Nausea (Gastrointestinal disorders) | 3
Rash (Skin and subcutaneous tissue disorders) | 1
Soreness at infusion site (Injury, poisoning and procedural complications) | 1
Vomiting (Gastrointestinal disorders) | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No